CLINICAL TRIAL: NCT04319965
Title: Complications Related to Transpulmonary Thermodilution in the Intensive Care Unit and the Operating Room
Brief Title: Complications Related to Transpulmonary Thermodilution
Acronym: COTRADIL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Xavier Monnet, Professor Xavier Monnet MD. PhD., Bicetre Hospital
Other Study IDs: 2018-A03234-51
Record Dates: First submitted 2020-03-13; First posted 2020-03-24 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Critical Illness; Hemodynamic Instability; Septic Shock; Acute Respiratory Distress Syndrome
Keywords: Hemodynamic monitoring; Transpulmonary Thermodilution; Intensive care unite; Operating room; Complications of catheters
MeSH Terms: conditions — Critical Illness; Shock, Septic; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The transpulmonary thermodilution is commonly used in patients with acute circulatory failure in the intensive care unit and for monitoring surgical patients at high risk. However, the incidence of complications and their risk factors in patients monitored by transpulmonary thermodilution has not been completely reported yet.

DETAILED DESCRIPTION:
Transpulmonary thermodilution (TPTD) is a technique used for haemodynamic monitoring. It consists of a monitor device which is connected to two catheters. One is a catheter inserted into the superior vena cava (internal jugular or subclavian), which is a standard catheter commonly used in patients with acute circulatory failure. The other one is a thermistor-tipped arterial catheter, which is inserted through the femoral route (the tip stands in the iliac artery), which allows the measurement of blood temperature. Catheters designed for the radial, brachial and humeral arteries also exist. TPTD allows the computation of cardiac output from the thermodilution curve recorded by the thermistor-tipped femoral arterial catheter. As an advanced cardiac output monitoring technique, it provides several important haemodynamic variables. It can be used in the intensive care unit (ICU) and in the operating room (OR). Two TPTD systems are now on the market. The PiCCO2 system (Pulsion Medical Systems, member of the Getinge Group, Feldkirchen, Germany) and the VolumeView/EV1000 system (Edwards Lifesciences, Irvine, United States of America). This study is designed to investigate the incidence of complications and their risk factors in patients monitored by transpulmonary thermodilution.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Monitoring by a TPTD system (PiCCO2 or VolumeView/EV1000) already planned or set up

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU or intermediate care units and in OR, monitoring by TPTD system
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-02-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
To describe the incidence of transpulmonary thermodilution related complications | At the time of TPTD catheters removal, an average of 7-14 days, depending on the individual situation
  Systematic report of mechanical, haemorragic and infections complications

SECONDARY OUTCOMES:
Prevalence of theoretical risk factors for these complications. | Through study completion, up to 1 year
  Systematic report of morphologic characteristics, coagulation, immunity

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Monnet, MD.PhD, Study Chair — Medical intensive care unit; Bicêtre Hospital
Locations (1):
- Bicetre Hospital, Paris, Val-de-Marne, France

REFERENCES:
- [Background] Sakka SG, Reuter DA, Perel A. The transpulmonary thermodilution technique. J Clin Monit Comput. 2012 Oct;26(5):347-53. doi: 10.1007/s10877-012-9378-5. Epub 2012 Jul 18. PMID 22806214
- [Background] Monnet X, Teboul JL. Transpulmonary thermodilution: advantages and limits. Crit Care. 2017 Jun 19;21(1):147. doi: 10.1186/s13054-017-1739-5. PMID 28625165
- [Background] Jozwiak M, Teboul JL, Monnet X. Extravascular lung water in critical care: recent advances and clinical applications. Ann Intensive Care. 2015 Dec;5(1):38. doi: 10.1186/s13613-015-0081-9. Epub 2015 Nov 6. PMID 26546321
- [Background] Vincent JL, Rhodes A, Perel A, Martin GS, Della Rocca G, Vallet B, Pinsky MR, Hofer CK, Teboul JL, de Boode WP, Scolletta S, Vieillard-Baron A, De Backer D, Walley KR, Maggiorini M, Singer M. Clinical review: Update on hemodynamic monitoring--a consensus of 16. Crit Care. 2011 Aug 18;15(4):229. doi: 10.1186/cc10291. PMID 21884645
- [Background] Cecconi M, De Backer D, Antonelli M, Beale R, Bakker J, Hofer C, Jaeschke R, Mebazaa A, Pinsky MR, Teboul JL, Vincent JL, Rhodes A. Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Dec;40(12):1795-815. doi: 10.1007/s00134-014-3525-z. Epub 2014 Nov 13. PMID 25392034
- [Background] Belda FJ, Aguilar G, Teboul JL, Pestana D, Redondo FJ, Malbrain M, Luis JC, Ramasco F, Umgelter A, Wendon J, Kirov M, Fernandez-Mondejar E; PICS Investigators Group. Complications related to less-invasive haemodynamic monitoring. Br J Anaesth. 2011 Apr;106(4):482-6. doi: 10.1093/bja/aeq377. Epub 2010 Dec 26. PMID 21205627